CLINICAL TRIAL: NCT02675569
Title: ACCESS HD Pilot: A Randomized Trial Comparing Catheters to Fistulas in Elderly patientS Starting HemoDialysis
Brief Title: ACCESS HD: Comparing Catheters to Fistulas in Elderly Patients Starting Hemodialysis
Acronym: ACCESS HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Applied Health Research Centre (Other); The George Institute (Other)
Responsible Party: Principal Investigator, Dr. Rob Quinn, Nephrologist and Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB14-1670
Record Dates: First submitted 2016-01-26; First posted 2016-02-05 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: End-stage Kidney Failure
Keywords: Vascular access; Hemodialysis; Kidney failure; Catheter; Fistula
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Fistula | interventions — Catheters; Portacaval Shunt, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter (Active Comparator): Catheter is a method of vascular access for hemodialysis. It consists of a long, thin plastic tube and may be either tunnelled or non-tunnelled.
  Interventions: Procedure: Catheter
- Fistula (Experimental): Fistula is a type of vascular access strategy for hemodialysis in which a direct connection of an artery to a vein is created. It is intended to provide an access with good blood flow that can last for decades.
  Interventions: Procedure: Fistula

INTERVENTIONS:
Procedure: Catheter — A method of vascular access for hemodialysis that all participants will have in place prior to randomization.
  Arms: Catheter
Procedure: Fistula — A type of vascular access strategy for hemodialysis which involves connecting the artery and the veins in the participant's arm.
  Arms: Fistula

SUMMARY:
This randomized controlled trial (RCT) is multi-center, parallel-arm, and open label. It will test the feasibility and safety of randomizing elderly patients with end-stage kidney failure starting hemodialysis with a tunneled/non-tunneled catheter to one of the following vascular access strategies: (a) attempt at fistula creation (intervention), or (b) continued use of a catheter (comparator). A total number of 100 participants will be enrolled in vanguard phase of the RCT. The rationale for this trial includes: (1) the importance of the intervention question related to the choice of vascular access for patients treated with hemodialysis; (2) lack of evidence from clinical trials for decision-making in this area (only observational studies are available); (3) existing studies which suggest that fistula use is associated with better patient outcomes are very prone to selection bias; (4) need for a clinical trial comparing the impact of the two most frequently chosen strategies for vascular access (catheter and fistula) in the hemodialysis population; and (5) a feasible and safe trial design. The results obtained from this vanguard phase of the RCT will determine the feasibility and safety of conducting a large RCT, which will be powered for the primary outcome of days spent in hospital.

DETAILED DESCRIPTION:
Purpose: This vanguard phase of the RCT will help to address challenges related to patient recruitment, protocol adherence, safety, and data collection in the hemodialysis population. The primary outcome for this vanguard phase of the RCT is feasibility, which will be measured by patient recruitment and protocol adherence. The secondary outcomes include feasibility-related outcomes, safety (which will include expected procedure-related outcomes and causes for hospital admissions), and other protocol violations.

Hypothesis: Results obtained from the vanguard phase of the RCT will provide feasibility and safety data for conducting a large RCT, which will establish a better understanding of the clinical outcomes associated with the use of fistula versus catheter for vascular access in the hemodialysis population.

Research Method: This is a multicenter, open-label, RCT, and is expected to be conducted over 24 months. All consented and enrolled participants who meet the eligibility criteria will have the following data collected in a minimal dataset: eligibility, age, sex, program/center, height, weight, comorbid conditions, and details of any prior treatment for acute or chronic kidney failure (e.g., previous peritoneal dialysis, kidney transplant, or hemodialysis). The following additional data will be collected at baseline: baseline laboratory values, baseline hemodialysis initiation, history of access procedures, and patient-reported outcome measures (includes data on quality of life and a vascular access questionnaire). The vanguard phase of the RCT will consist of 6 months of site preparation, approximately 24 months of participant accrual, and 6 months of additional follow-up time for the last randomized participant. An additional 6 months will be used to assess the preliminary data, prepare the report of this vanguard phase of the RCT, and to prepare and submit funding applications for the large RCT. Participants in the vanguard phase of the RCT will be rolled into the large RCT, and will therefore be followed for a total of 24 months (2 years) in Canada and a total of 36 months (3 years) in Australia after randomization to assess adherence to the trial protocol, assess safety outcomes, and collect qualitative data.

Statistical Analysis Plan: The primary analysis of the vanguard phase of the RCT will be descriptive. The proportion of people meeting each of the feasibility endpoints with accompanying 95% confidence intervals will be calculated. Investigators will describe participant characteristics and evaluate reasons for protocol violation, as well as calculate rates of drop-ins and other events. Interim or subgroup analyses will not be conducted in this vanguard phase of the RCT.

Expected Procedure-Related Outcomes (Safety Data): As both catheter and fistula treatment strategies are standard of care, the procedure-related outcomes are well known. Investigators will collect only expected procedure-related outcomes (i.e., events that have a potentially causal relationship to the strategy) that occur within 7 days of the execution of any access related intervention. These will include hospital admissions and prolongation of hospitalization, status changes, bacterial infections, catheter or exit site infections, cannulation injury events. In addition, sites will report all incidents of participant death that occur during the trial period. Cause of death will be determined by trial site investigators, based on a trial-specific list of classifications, and will be adjudicated for accuracy by appropriate members of the trial steering committee, who will be blinded to treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age ≥ 55; (AUS sites : adult patients age ≥ 65);
2. a). Started hemodialysis using a tunnelled, or non-tunnelled catheter for vascular access AND ≤ 1 previously unsuccessful fistula attempt; OR b).Changing over from peritoneal dialysis AND no functioning arteriovenous fistula available at HD start;
3. Treated with hemodialysis for 365 days or less at the time of consent (374 days or less at the time of randomization);
4. Clinically and cognitively stable (able to provide consent within 365 days of hemodialysis start);
5. Hemodialysis is the intended modality of treatment;
6. End-stage (permanent) kidney failure unlikely to recover kidney function according to the attending nephrologist;
7. Eligible for a fistula attempt as determined by the local multidisciplinary access team;
8. Planning to remain in the current dialysis center/service for at least 6 months;

Exclusion Criteria:

1. Started hemodialysis with a fistula or have a patent fistula already in place or had >1 unsuccessful attempt; (AUS sites: or previously functioning fistula no longer working);
2. . Has had a prior arteriovenous graft creation;
3. Imminent transplant planned (within 6 months);
4. Metastatic malignancy or other condition associated with a life expectancy of less than 6 months, in the opinion of the attending nephrologist;

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility; proportion of eligible people who are randomized (at least 25%) | 42 months
Feasibility; proportion of those randomized to the intervention arm receiving a fistula attempt within 90 days of randomization (at least 80%) | 42 months

SECONDARY OUTCOMES:
Descriptive; reasons for exclusion of all screened participants (feasibility) | 42 months
  Investigators will consider the reasons for exclusion of screened participants (including competing studies).
Descriptive; reasons that people decline to participate (feasibility) | 42 months
  Investigators will consider the reasons that people decline to participate.
Descriptive; reasons people are considered ineligible for a fistula attempt (feasibility) | 42 months
  Investigators will consider the reasons that people are considered ineligible for a fistula attempt.
Descriptive; reasons for delayed access to fistula surgery (feasibility) | 42 months
  Investigators will consider the reasons for delayed access to fistula surgery (> 90 days from randomization).
Safety; expected procedure-related outcomes for both catheter and fistula treatment strategies that occur within 7 days of the execution of any access related intervention | 7 days
  Investigators will collect information on expected procedure-related outcomes for both catheter and fistula treatment strategies that occur within 7 days of the execution of any access related intervention. Additionally, coordinators will track causes for hospital admissions and prolongation of hospitalization, and sites will report all incidents of participant death that occur during the trial period to identify if outcomes may have resulted from the trial procedures.
Number of drop-ins | 42 months
  Investigators will collect the number and reasons for drop-ins and drop-outs.
Number of drop-outs | 42 months
  Investigators will collect the number and reasons for drop-ins and drop-outs.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Quinn, PhD, Principal Investigator — University of Calgary; Pietro Ravani, PhD, Principal Investigator — University of Calgary
Locations (13):
- Australia (3):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Illawarra Shoalhaven Local Health District (ISLHD), Wollongong, New South Wales
  - Sunshine Coast Hospital and Health Service (SCHHS), Birtinya, Queensland
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - St. Joseph's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee H, Manns B, Taub K, Ghali WA, Dean S, Johnson D, Donaldson C. Cost analysis of ongoing care of patients with end-stage renal disease: the impact of dialysis modality and dialysis access. Am J Kidney Dis. 2002 Sep;40(3):611-22. doi: 10.1053/ajkd.2002.34924. PMID 12200814
- [Background] Jindal K, Chan CT, Deziel C, Hirsch D, Soroka SD, Tonelli M, Culleton BF; Canadian Society of Nephrology Committee for Clinical Practice Guidelines. Hemodialysis clinical practice guidelines for the Canadian Society of Nephrology. J Am Soc Nephrol. 2006 Mar;17(3 Suppl 1):S1-27. doi: 10.1681/ASN.2005121372. No abstract available. PMID 16497879
- [Background] Ravani P, Palmer SC, Oliver MJ, Quinn RR, MacRae JM, Tai DJ, Pannu NI, Thomas C, Hemmelgarn BR, Craig JC, Manns B, Tonelli M, Strippoli GF, James MT. Associations between hemodialysis access type and clinical outcomes: a systematic review. J Am Soc Nephrol. 2013 Feb;24(3):465-73. doi: 10.1681/ASN.2012070643. Epub 2013 Feb 21. PMID 23431075
- [Background] Quinn RR, Laupacis A, Hux JE, Oliver MJ, Austin PC. Predicting the risk of 1-year mortality in incident dialysis patients: accounting for case-mix severity in studies using administrative data. Med Care. 2011 Mar;49(3):257-66. doi: 10.1097/MLR.0b013e318202aa0b. PMID 21301370
- [Background] Tennankore KK, Soroka SD, Kiberd BA. The impact of an "acute dialysis start" on the mortality attributed to the use of central venous catheters: a retrospective cohort study. BMC Nephrol. 2012 Jul 30;13:72. doi: 10.1186/1471-2369-13-72. PMID 22846341
- [Background] Mazonakis E, Stirling C, Booth KL, McClenahan J, Heron N, Geddes CC. The influence of comorbidity on the risk of access-related bacteremia in chronic hemodialysis patients. Hemodial Int. 2009 Jan;13(1):6-10. doi: 10.1111/j.1542-4758.2009.00327.x. PMID 19210271
- [Background] Lok CE, Allon M, Moist L, Oliver MJ, Shah H, Zimmerman D. Risk equation determining unsuccessful cannulation events and failure to maturation in arteriovenous fistulas (REDUCE FTM I). J Am Soc Nephrol. 2006 Nov;17(11):3204-12. doi: 10.1681/ASN.2006030190. Epub 2006 Sep 20. PMID 16988062
- [Background] Quinn RR, Lamping DL, Lok CE, Meyer RA, Hiller JA, Lee J, Richardson EP, Kiss A, Oliver MJ. The Vascular Access Questionnaire: assessing patient-reported views of vascular access. J Vasc Access. 2008 Apr-Jun;9(2):122-8. PMID 18609528
- [Background] Oliver MJ, Verrelli M, Zacharias JM, Blake PG, Garg AX, Johnson JF, Pandeya S, Perl J, Kiss AJ, Quinn RR. Choosing peritoneal dialysis reduces the risk of invasive access interventions. Nephrol Dial Transplant. 2012 Feb;27(2):810-6. doi: 10.1093/ndt/gfr289. Epub 2011 Jun 21. PMID 21693682
- [Background] Tordoir J, Canaud B, Haage P, Konner K, Basci A, Fouque D, Kooman J, Martin-Malo A, Pedrini L, Pizzarelli F, Tattersall J, Vennegoor M, Wanner C, ter Wee P, Vanholder R. EBPG on Vascular Access. Nephrol Dial Transplant. 2007 May;22 Suppl 2:ii88-117. doi: 10.1093/ndt/gfm021. No abstract available. PMID 17507428
- [Background] Casey JR, Hanson CS, Winkelmayer WC, Craig JC, Palmer S, Strippoli GF, Tong A. Patients' perspectives on hemodialysis vascular access: a systematic review of qualitative studies. Am J Kidney Dis. 2014 Dec;64(6):937-53. doi: 10.1053/j.ajkd.2014.06.024. Epub 2014 Aug 10. PMID 25115617
- [Background] Detry MA, Lewis RJ. The intention-to-treat principle: how to assess the true effect of choosing a medical treatment. JAMA. 2014 Jul 2;312(1):85-6. doi: 10.1001/jama.2014.7523. No abstract available. PMID 25058221
- [Background] Murea M, James KM, Russell GB, Byrum GV 3rd, Yates JE, Tuttle NS, Bleyer AJ, Burkart JM, Freedman BI. Risk of catheter-related bloodstream infection in elderly patients on hemodialysis. Clin J Am Soc Nephrol. 2014 Apr;9(4):764-70. doi: 10.2215/CJN.07710713. Epub 2014 Mar 20. PMID 24651074
- [Derived] Quinn R, Ravani P; ACCESS HD Investigators. ACCESS HD pilot: A randomised feasibility trial Comparing Catheters with fistulas in Elderly patientS Starting haemodialysis. BMJ Open. 2016 Nov 24;6(11):e013081. doi: 10.1136/bmjopen-2016-013081. PMID 27884849